CLINICAL TRIAL: NCT06895538
Title: An Exploratory, Non-Randomized, Controlled Study of the Effect of Rabbit Anti-Human T-Lymphocyte Immunoglobulin (ATLG) Versus Anti-Thymocyte Immunoglobulin (ATG) on Immune Reconstitution After Allogeneic Hematopoietic Stem Cell Transplantation for Malignant Hematologic Diseases
Brief Title: Comparison of ATLG and ATG for Immune Reconstitution After Allo-HSCT for Hematologic Malignancy
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKUFH 2024 644-002
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Leukemia; MDS; Lymphoma
Keywords: ATLG; ATG; immune reconstitution; allo-HSCT
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anti-human T-lymphocyte rabbit immunoglobulin (ATLG): ATLG will be given as a substitute for ATG in the conditioning regimen for hematologic malignancy patients who are undergoing allo-HSCT
  Interventions: Drug: Rabbit Anti-Human T-Lymphocyte Immunoglobulin (ATLG)

INTERVENTIONS:
Drug: Rabbit Anti-Human T-Lymphocyte Immunoglobulin (ATLG) — Patients in the ATLG arm receive ATLG instead of ATG as part of the routine conditioning regimen before allo-HSCT; ATLG is given intravenously by infusion for 4 consecutive days, after which they undergo routine transplantation.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation is the only curative treatment for malignant hematologic diseases. However, immune rejection is a major limitation in its application. In the "Beijing Protocol", the use of granulocyte colony-stimulating factor (G-CSF) in combination with anti-thymocyte globulin (ATG) can achieve "everyone has a donor". The use of ATG, however, can interfere with the recovery of immune function after transplantation, increasing the risk of life-threatening complications such as viral infections or graft-versus-host disease. Rabbit anti-human T-lymphocyte immunoglobulin (ATLG) is currently approved for the prevention of organ transplant rejection, which is produced differently from ATG. Previous studies have shown that transplant preconditioning with ATLG is effective in preventing graft-versus-host disease and even reduces the incidence of cytomegalovirus, etc. after transplantation. In this study, we will prospectively apply containing ATLG in a cohort of allogeneic hematopoietic stem cell transplantation for malignant hematologic diseases and dynamically observe the state of immune reconstitution of patients after transplantation. We will also compare it with a matched cohort of conventional combined ATGs during the same period to explore the impact of ATLG on immune reconstitution after transplantation.

DETAILED DESCRIPTION:
Hematological malignancies (referred to as malignant hematological diseases) are a class of major diseases that pose a significant threat to human health. Currently, allogeneic hematopoietic stem cell transplantation (allo-HSCT) remains an effective, if not the sole, treatment option for hematological tumors. Due to the potential for immune rejection, HSCT has historically been constrained to HLA-compatible siblings or non-consanguineous donors, significantly restricting its clinical application. In consideration of the findings from preceding studies, Huang's research team employed the immunomodulatory property of G-CSF in conjunction with anti-thymocyte globulin (ATG) to undertake the non-in vitro eradication of T lymphocytes for haplotype-conjugate HSCT. A series of studies were published in 2004 and 2013 that utilized G-CSF in combination with ATG to facilitate HSCT implantation. These studies demonstrated a correlation between the degree of HLA non-conformity and the degree of graft-versus-host disease (GVHD). This suggests that G-CSF combined with ATG successfully crosses the human leukocyte antigen (HLA) barrier, and that haploidentical transplantation has gradually become the most clinically utilized type of transplantation. However, clinical studies and real-world results have demonstrated that the application of ATG has the potential to enhance the risk of post-transplant cytomegalovirus (CMV), EBV activation or even infection, and post-transplant lymphoproliferative disease (PTLD).

A study published in 2023 utilized a retrospective analysis of clinical outcomes to examine patients who received two distinct sources of allogeneic T-cell-depleted (ATG) transplants. The findings indicated that patients who received ATLG during transplantation exhibited a reduced incidence of cytomegalovirus (CMV) infection. In a seminal study, Wang Shunqing and colleagues investigated the role, toxicities, and effects of ATG/ATLG on transplantation complications in non-myeloablative hematopoietic stem cell transplantation. Their findings demonstrated that the administration of ATG/ATLG during non-myeloablative hematopoietic stem cell transplantation was both safe and effective. Notably, it was observed to promote the implantation of hematopoietic stem cells, reduce the incidence of acute graft-versus-host disease (aGVHD), and decrease its severity. Huang Wenrong and colleagues investigated the effectiveness and safety of ATLG/ATLG in unrelated donor allogeneic peripheral hematopoietic stem cell transplantation. The study demonstrated that ATLG significantly reduced the incidence of cGVHD, decreased the occurrence of adverse events, and effectively controlled the occurrence of aGVHD. Lu Daopei et al. investigated the effectiveness and safety of ATG/ATLG in haploidentical hematopoietic stem cell transplantation to prevent graft-versus-host disease (GVHD). Their findings indicated that the dosage of ATG, at 7.5 mg/kg, was equivalent to the dosage of ATLG, at 20 mg/kg, in the context of haploidentical hematopoietic stem cell transplantation. Consequently, ATLG has been extensively utilized for immunosuppressive therapy in patients with hematologic disorders undergoing hematopoietic stem cell transplantation.

A paucity of studies currently exists on the effect of ATLG on immune reconstruction after HSCT and on comparison with ATG treatment modalities. The objective of this study is to prospectively apply ATLG pretreatment in a cohort of allogeneic HSCT for malignant hematologic diseases. The study will dynamically observe the status of immune reconstruction in post-transplantation patients and compare it with a cohort of conventional combined ATG during the same period. The primary research question guiding this study is to explore the effect of ATLG on immune reconstitution after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 1）Age ≧18 years, gender is not limited;
* 2）Histologically or cytologically confirmed diagnosis of malignant hematologic diseases;
* 3) First time undergoing allogeneic hematopoietic stem cell transplantation;
* 4) ECOG score 0-2;
* 5) Hepatic and renal function, cardiopulmonary function meet the following requirements.

  * Serum creatinine ≤ 1.5 ULN; ②Left ventricular ejection fraction ≥ 45%;

    * Blood oxygen saturation >91%;

      * Total bilirubin ≤ 2 × ULN; ALT and AST ≤ 3 × ULN; for ALT and AST abnormalities due to disease (e.g., liver infiltrates or bile duct obstruction), in the judgment of the investigator, the values may be adjusted to ≤ 5 × ULN;
* 6) Expected survival is longer than 12 weeks;
* 7) The subjects will voluntarily and strictly comply with the requirements of the study protocol and will sign a written informed consent form.

Exclusion Criteria:

* 1) Prior treatment with ATG, ALG, or ATLG drugs within the past six months;
* 2) Allergic to any component of ATLG or ATG;
* 3) Bacterial, viral, parasitic, or mycobacterial infections not adequately controlled by treatment, i.e., inability to undergo hematopoietic stem cell transplantation due to severe infection.

  4) Women who are pregnant or breastfeeding, or participants of childbearing potential who are unwilling or unable to use effective methods of contraception; 5) Participants enrolled in another clinical trial (of any investigational drug or device) within 30 days prior to the subject's baseline visit. (Subjects enrolled in observational studies are eligible to participate).

  6) Any other circumstance that, in the judgment of the investigator, may interfere with the conduct of the clinical trial and the determination of the results of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of hematologic malignancy undergoing allogeneic hematopoietic stem cell transplantation at Peking University First Hospital will be invited to participate in the study if they meet the enrollment criteria and are fully informed.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-05-03 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of viral infections after hematopoietic stem cell transplantation | From enrollment to 1 year after allo-HSCT
  Incidence of CMV reactivation (CMV DNA ≥10^3) and CMV disease, incidence of EBV reactivation (incidence of EBV DNA ≥10^5) and lymphoproliferative disorders (PTLD), incidence of hemorrhagic cystitis, incidence of herpes simplex, adenovirus, or other viruses in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
Not decided